CLINICAL TRIAL: NCT01631968
Title: Incidence of Infection After Total Knee Arthroplasty Using an Erythromycin and Colistin Loaded Cement or a Standard Cement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Pedro Hinarejos, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERITR-COL
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2012-06

CONDITIONS: Infection After Primary Total Knee Arthroplasty
MeSH Terms: interventions — Dental Cements; Anti-Bacterial Agents; Colistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cement with erytromycin and colistin (Experimental): In this group the knee arthroplasty was fixed with cement with erythromycin and colistin.
  Interventions: Procedure: Cement with erytromycin and colistin.
- Cement without antibiotic (Placebo Comparator): In this group the knee arthroplasty was fixed with standard cement, without any antibiotics.
  Interventions: Procedure: Cement without antibiotic.

INTERVENTIONS:
Procedure: Cement without antibiotic.
  Arms: Cement without antibiotic
Procedure: Cement with erytromycin and colistin.
  Arms: Cement with erytromycin and colistin

SUMMARY:
Prospective randomized study in cemented primary total knee arthroplasty. In one group the cement used was standard cement, without any antibiotics and in the other group the cement used was loaded with 0.5 g of erythromycin and 3 million units of colistin in 40 g of cement. In all cases intravenous antibiotics prophylaxis against infection was used. In both groups the cement was mechanically mixed in a vacuum. One deep drain tube was placed for 24 hours in all cases. The main variable was the presence of infection according to the Center of Disease Control criteria with a minimum of 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Primary total knee replacement. Both genders. No age limits.

Exclusion Criteria:

* Allergy to erythromycin or colistin. Previous infection in the knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2948 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Infection | The minimum follow-up is 12 months.
  Presence or absence of infection, according to the Center for Disease Control's criteria. The infection cases are classified as superficial of deep infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Esperanza., Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Hinarejos P, Guirro P, Leal J, Montserrat F, Pelfort X, Sorli ML, Horcajada JP, Puig L. The use of erythromycin and colistin-loaded cement in total knee arthroplasty does not reduce the incidence of infection: a prospective randomized study in 3000 knees. J Bone Joint Surg Am. 2013 May 1;95(9):769-74. doi: 10.2106/JBJS.L.00901. PMID 23636182